CLINICAL TRIAL: NCT05659563
Title: Preoperative Window of Opportunity Study With Giredestrant (GDC-9545) or Tamoxifen in Premenopausal Women With Estrogen Receptor-Positive/Human Epidermal Growth Factor Receptor 2-Negative & Ki67≥10% Early Breast Cancer
Brief Title: Preoperative Window Opportunity Study With Giredestrant or Tamoxifen in Premenopausal Women With ER+/HER2[-] & Ki67≥10%
Acronym: EMPRESS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEDOPP459; 2022-002166-33 (EudraCT Number); 2023-503565-36-00 (Other: EU CT Number)
Record Dates: First submitted 2022-12-05; First posted 2022-12-21 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Breast Cancer, Early-Onset
MeSH Terms: conditions — Breast Neoplasms | interventions — giredestrant; Tamoxifen

STUDY DESIGN:
Intervention Model Description: Multicenter, international, open-label, two-arms, one stage, phase II, window of opportunity, clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Giredestrant (GDC-9545): 30mg, orally (PO), daily (QD) during 15 days
  Interventions: Drug: Giredestrant
- Arm B (Active Comparator): Tamoxifen: 20mg, orally (PO), daily (QD) during 15 days
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Giredestrant — Giredestrant is a highly potent, non-steroidal, oral selective ER antagonist and degrader (SERD)
  Other Names: GDC-9545
  Arms: Arm A
Drug: Tamoxifen — Tamoxifen is a selective estrogen receptor (ER) modulator
  Other Names: Nolvadex® or Soltamox®
  Arms: Arm B

SUMMARY:
This study is a window of opportunity clinical trial to evaluate the efficacy of giredestrant (GDC-9545) or tamoxifen in estrogen receptor-positive (ER[+])/human epidermal growth factor receptor 2-negative (HER2[-]) primary invasive adenocarcinoma of the breast with Ki67 level ≥ 10%.

A total of 92 patients will be enrolled in this trial and randomized 1:1 in the arm A with giredestrant (GDC-9545) and the arm B with tamoxifen, with a total duration of treatment of 15 days.

This study will analyze the efficacy of giredestrant (GDC-9545) as determined by Ki67 expression between baseline tumor biopsy samples and post-treatment biopsy samples.

DETAILED DESCRIPTION:
This is a multicenter, international, open-label, two-arms, one stage, phase II, preoperative window of opportunity clinical trial to evaluate the efficacy of giredestrant (GDC-9545) as single agent in ER[+]/HER2[-] early breast cancer patients with Ki67 ≥ 10%.

Upon meeting all selection criteria, 92 patients enrolled in the study will receive either giredestrant (GDC-9545) 30 mg or tamoxifen .

A total of 92 patients will be enrolled as follows:

* 46 patients in the investigational Arm A will receive giredestrant [GDC-9545] 30 mg. It will be administered orally once a day during 15 days.
* 46 patients in the control Arm B will receive tamoxifen 20 mg. It will be administered orally once a day during 15 days.

Patients can take both treatments at home.

The main objective is to analyze the efficacy of giredestrant (GDC-9545) according to changes in tumor cell proliferation. This analysis will compare absolute changes for Ki67 expression between baseline score and the evaluation after 15 days of treatment.

Total study duration is 15 days of treatment and until 28 days after the last dose of the study treatment (or discontinuation) of follow up.

ELIGIBILITY:
Inclusion criteria

Patients must meet ALL the following inclusion criteria to be eligible for enrolment into the study:

1. Signed Informed Consent Form (ICF) prior to beginning specific protocol procedures.
2. Aged ≥ 18 years at time of signing ICF.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Women in a well-determined premenopausal status as indicated in the protocol Section 4.1.
5. Histologically confirmed invasive breast carcinoma, with all the following characteristics:

   1. Documented ER-positive tumor in accordance with American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines (Allison et al., 2020), assessed locally and defined as ≥ 1% of tumor cells stained positive.
   2. Documented HER2-negative tumor in accordance with 2018 ASCO/CAP guidelines (Wolff et al., 2018), assessed locally at baseline.

      Note: Diagnostic biopsy taken no more than 8 weeks prior to initiation of study treatment can be used as baseline.
   3. Ki67 score ≥10% analyzed locally and centrally confirmed (Nielsen et al., 2021).

      Note: Ki67 will be analyzed locally at the time of inclusion. Patients with basal Ki67 ≥20% will be assessed locally and centrally confirmed retrospectively and patients with 10-19% will be assessed centrally before inclusion.
   4. Tumor size must be ≥1.0 cm in longest diameter by ultrasound as per Response Evaluation Criteria in solid Tumors (RECIST) criteria.

   Note: Patients with multifocal or multicentric breast cancer with a at least one tumor lesion ≥1.0 cm in the longest diameter by ultrasound (reference lesion) are also eligible if the two largest lesions have been histologically confirmed in the clinical evaluation and meet pathologic criteria for ER positivity and HER2 negativity.
6. Willingness to provide a primary tumor tissue and blood sample obtained at baseline as well as a post-treatment tumor tissue and blood samples (breast biopsy or from breast surgery).
7. Patient has adequate bone marrow, liver, and renal function:

Hematological: absolute neutrophil count (ANC) ≥ 1.5 x 109/L (1500/mL), platelet count ≥ 100.0 x109/L, and hemoglobin ≥ 9 g/dL (≥ 90g/L).

Note: The blood counts are to meet the specified criteria without transfusion or growth factor support, unless it is clear that the bone marrow function is adequate and that any aberration has a clear and correctable cause, and the correction undertaken.

Hepatic: total serum bilirubin ≤ 1.5' institutional upper limit of normal (ULN) (patients with known Gilbert's syndrome: ≤ 3' ULN); alkaline phosphatase (ALP) ≤ 2.5 times ULN; aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤ 3' times ULN.

Coagulation: The international normalized ratio (INR) < 1.5' ULN and partial thromboplastin time (PTT or aPTT) < 1.5' ULN (except for patients receiving anticoagulation therapy). For patients receiving warfarin, a stable INR between 2 and 3 is required. For patients receiving heparin, PTT (or aPTT) between 1.5 and 2.5' ULN (or patient value before starting heparin treatment) is required. If anticoagulation therapy is required for a prosthetic heart valve, stable INR between 2.5 and 3.5 is permitted.

Renal: creatinine clearance ≥ 60 mL/min for patients with creatinine levels above institutional normal.

Negative serum pregnancy test result within 14 days prior to initiation of study treatment and a negative urine pregnancy test within 24 hours prior to study treatment initiation.

Note: Premenopausal women age ≥18 years with premenopausal status defined as: estradiol (E2) in the premenopausal range (according to institution parameters) or patient has been menstruating regularly during the 6 months prior to randomization and has not used any form of hormonal contraception or any other hormonal treatments during this time.

Women must remain abstinent and truly abstains from sexual activity (refrains from heterosexual intercourse) or use of locally recognized adequate methods of contraception (described as that with a failure rate <1%) during the length of the study, and to continue its use for 10 days after the last dose of study treatment (for patients taking giredestrant) or 9 months following cessation of therapy (for patients in the tamoxifen arm). They must, as well, agree to refrain from donating eggs during the same period of time.

Examples of non-hormonal contraceptive method with a failure rate of <1% per year (e.g. bilateral tubal ligation, male sterilization and copper intrauterine devices). The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the individual. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception.

9. Patients must be accessible for treatment and follow-up.

10. Participants who are able and willing to swallow, retain, and absorb oral medication.

Exclusion criteria

1. Patients will be excluded from the study if they meet ANY of the following criteria:
2. Progesterone receptor (PgR)[+] and ER[-] patients.

   cT4 and/or cN2/3 and/or bilateral BC.
3. Patients who have history of any prior (ipsilateral and/or contralateral) invasive BC or Ductal carcinoma in situ (DCIS). Participants with a history of contralateral DCIS treated by only local regional therapy at any time may be eligible.
4. Evidence of metastatic disease.
5. Previous systemic or local treatment for the primary BC currently under investigation.
6. History of any prior treatment with chemotherapy drugs, aromatase inhibitors (AIs), tamoxifen, selective estrogen receptor down regulator, or cyclin-dependent kinase 4 and 6 inhibitors (CDK4/6i).
7. Any invasive malignancy diagnosed within the previous 5 years prior to screening in this study (other than basal cell carcinoma, cervical carcinoma in situ or contralateral DCIS).
8. Known issues with swallowing oral medication, or inability or unwillingness to swallow oral medication.
9. Participants who have a known clinically significant history of liver disease consistent with Child-Pugh Class B or C, including hepatitis (e.g., hepatitis B virus [HBV] or hepatitis C virus [HCV]), current alcohol abuse, cirrhosis, or positive test for viral hepatitis, as defined below:
10. Active infection is defined as requiring treatment with antiviral therapy or presence of positive test results for hepatitis B (hepatitis B surface antigen and/or total hepatitis B core antibody [HBcAb]) or HCV antibody. Unless required by local regulations, participants are not required to have HBV, or HCV assessments at screening if these assessments have not been previously performed.

    Participants who test positive for HBcAb are eligible only if test results are also positive for hepatitis B surface antibody and polymerase chain reaction is negative for HBV DNA Participants who are positive for HCV serology are eligible only if testing for HCV RNA is negative.

    Active cardiac disease or history of cardiac dysfunction including any of the following:

    History or presence of symptomatic bradycardia or sick sinus syndrome.

    Resting heart rate < 50 bpm at screening.

    History of angina pectoris, symptomatic pericarditis, myocardial infarction, or any cardiac arrhythmias (e.g.,ventricular, supraventricular, nodal arrhythmias, or conduction abnormality) within 12 months prior to study entry.

    History of documented congestive heart failure (New York Heart Association Class II-IV) or cardiomyopathy.

    QT interval corrected through use of Fridericia's formula (QTcF) >470 ms by at least three ECGs >30 minutes apart.

    History of long or short QT syndrome, Brugada syndrome or known history of corrected QT interval prolongation, or torsades de pointes.

    History or presence of an abnormal ECG that is clinically significant in the investigator's opinion.

    History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias such as structural heart disease (e.g., severe left ventricular systolic dysfunction, left ventricular hypertrophic cardiomyopathy, infiltrative cardiomyopathy, moderate-to-severe valve disease), coronary heart disease (symptomatic or with ischemia demonstrated by diagnostic testing), clinically significant electrolyte abnormalities (e.g., hypokalemia, hypomagnesemia, hypocalcemia), or family history of long QT syndrome.
11. Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study.
12. Treatment with strong CYP3A4 inhibitors or inducers within 14 days or 5 drug elimination half-lives (whichever is longer) prior to randomization.
13. Active inflammatory bowel disease or chronic diarrhea, short bowel syndrome, or major upper gastrointestinal surgery including gastric resection.
14. Participants who have a known allergy or hypersensitivity to any of the study drugs or any of their excipients.
15. Participants who are pregnant or breastfeeding or intending to become pregnant during the study or within 10 days after the final dose of giredestrant (GDC-9545), or within 9 months after the final dose of tamoxifen.

    Note: Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment and a negative urine pregnancy test within 24 hours prior to study treatment initiation.
16. Patients with renal dysfunction who require dialysis.
17. Participants who have had a serious infection requiring oral or IV antibiotics within 14 days prior to screening or other clinically significant infection (e.g., COVID-19) within 14 days prior to screening.

    Note: Participants who have fully recovered from serious or clinically significant infections at least 14 days prior to screening are eligible. If a participant exhibits signs or symptoms of potential COVID-19 infection and there is a reasonable suspicion of exposure, investigators are to follow the American Society of Clinical Oncology 2020 guidelines or institutional guidelines on testing.
18. Participants who have had a major surgical procedure unrelated to breast cancer within 28 days prior to randomization.
19. Participants who are unable or unwilling to comply with the requirements of the protocol in the opinion of the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Change in proliferative index (Ki67 expression) | Baseline up to 15 days
  To assess changes in tumor cell proliferation as measured by Ki67 expression between baseline and D15 (+1 day) post-treatment tumor biopsy samples by central assessment in patients with centrally confirmed Ki67 ≥10% (Arm A: giredestrant vs Arm B: tamoxifen)

SECONDARY OUTCOMES:
Complete cell cycle arrest (CCCA) | Baseline up to 15 days
  To measure complete cell cycle arrest in all arms, defined as the percentage of participants with centrally assessed Ki67 scores ≤2.7% stained nuclei upon treatment
Changes in molecular profiles of tumor tissue samples | Baseline up to 15 days
  To analyze gene expression profiles in tumor tissue samples obtained at baseline and after treatment using the HTG EdgeSeq Oncology Biomarker Panel
Changes in expression levels of estrogen receptor and progesterone receptor in tumor tissue samples | Baseline up to 15 days
  To analyze the expression of estrogen receptor and progesterone receptor in tumor tissue samples obtained at baseline and post-therapy

OTHER OUTCOMES:
Changes in molecular profiles of plasma biomarkers related to endocrine function | Baseline up to 15 days
  To compare the expression of blood biomarkers in samples obtained at baseline and post-therapy using a plasma endocrine panel
Incidence and severity of adverse events | Baseline up to 15 days
  To evaluate incidence and severity of adverse events, with severity determined in accordance to NCI-CTCAE v.5.0

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Llombart, MD, Principal Investigator — Arnau de Vilanova Hospital, Valencia (Spain)
Locations (18):
- France (2):
  - Hopital Europeen Georges Pompidou, Paris
  - Hôpital Tenon AP-HP, Paris
- Spain (16):
  - Institut Català d' Oncologia Badalona, Badalona, Barcelona
  - Hospital Universitari Sant Joan de Reus, Reus, Tarragona
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Universitari Dexeus, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Clínico San Cecilio de Granada, Granada
  - Hospital Universitario de León, León
  - Hospital Beata Maria Ana, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Arnau de Vilanova de Valencia, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Instituto Valenciano de Oncología, Valencia

IPD SHARING:
Plan to Share IPD: No